CLINICAL TRIAL: NCT03819101
Title: A Phase III Trial of Acetylsalicylic Acid and Atorvastatin in Patients With Castrate-resistant Prostate Cancer
Brief Title: Trial of Acetylsalicylic Acid and Atorvastatin in Patients With Castrate-resistant Prostate Cancer
Acronym: PEACE-4
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2017-004639-35; 2017/2601 (Other: CSET number)
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Aspirin; Atorvastatin

STUDY DESIGN:
Intervention Model Description: This is a 2x2 factorial randomized, multicenter, international, open phase III trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A (No Intervention): Standard of Care (SOC) for CRPC
- Arm B (Experimental): SOC + acetylsalicylic acid 100 mg daily
  Interventions: Drug: Acetylsalicylic acid
- Arm C (Experimental): SOC + atorvastatin 80 mg daily
  Interventions: Drug: Atorvastatin
- Arm D (Experimental): SOC + acetylsalicylic acid 100 mg daily + atorvastatin 8
  Interventions: Drug: Acetylsalicylic acid; Drug: Atorvastatin

INTERVENTIONS:
Drug: Acetylsalicylic acid — 100mg
  Arms: Arm B; Arm D
Drug: Atorvastatin — 80 mg
  Arms: Arm C; Arm D

SUMMARY:
This is a 2x2 factorial randomized, multicenter, international, open phase III trial.

The primary objective is to evaluate the benefit of acetylsalicylic acid and atorvastatin on overall survival (OS) (main endpoint) for patients with castrate-resistant prostate cancer starting first line treatment for CRPC

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate and no curative local therapy considered possible
* Age ≥ 18 years, life expectancy of at least 6 months
* CRPC defined as tumor progression (PSA increase on at least 2 separate values separated by at least 1 week or progression on imaging) while on Androgen Deprivation Therapy (orchiectomy, LHRH agonist or -antagonist) with documented serum testosterone levels ≤ 1.7 nmol/L (≤ 0.50 ng/mL). Ongoing concurrent use of LHRH agonist or antagonist is required if the patient has not been surgically castrated
* Presence (M1) or absence (M0) of metastases on imaging
* Performance status 0, 1 or 2
* No previous use of life- prolonging treatments for CRPC (including abiraterone, enzalutamide, radium-223, docetaxel, cabazitaxel, and sipuleucel-T). The use of these agents together with Androgen Deprivation Therapy (ADT) for castrate-sensitive disease is allowed.
* Adequate renal function within 30 days prior to registration: calculated creatinine clearance ≥ 50 mL/min, according to the formula of Cockcroft-Gault and adequate liver function with levels of AST and ALT ≤ 3xULN and no signs for cholestasis.
* Participation in other clinical trials is allowed except for trials with the same primary endpoint, i.e. OS
* Patient authorized to participate to a clinical trial by specific country regulation (eg patient affiliated to a social security system or beneficiary of the same)
* Information delivered to patient and informed consent form signed by the patient.

Exclusion Criteria:

* Previous localised malignancy within 2 years with the exception of localized non-melanoma skin cancer and Ta or Tis bladder cancer (patients with asymptomatic Chronic Lymphocytic Leukemia can be included)
* Previous metastatic malignancy within 5 years
* Patient currently taking daily acetylsalicylic acid or a daily statin within the last 6 months
* Patients with active liver disease (hepatitis B or C, cirrhosis) or unexplained persistent elevations of serum transaminases exceeding 3 times the upper limit of normal or cholestasis
* Patients with excessive alcohol intake or history of a relevant liver disease
* Known hypersensitivity or intolerance to acetylsalicylic acid or atorvastatin or hypersensitivity to any of its components
* Contra-indication to acetylsalicylic acid or atorvastatin according to label, including known high-risk for haemorrhage,
* History of or active myopathy or significantly elevated (> 5 times ULN) CK levels
* History of recent stroke or transient ischemic attack (TIA).
* Any concomitant drugs contraindicated for use with the trial drugs according to the product information (e.g. Fusidic acid, potent inhibitors of CYP3A4 or transport proteins: ciclosporin, telithromycin, clarithromycin, delavirdine, stiripentol, ketoconazole, voriconazole, itraconazole, posaconazole and HIV protease inhibitors including ritonavir, lopinavir, atazanavir, indinavir, darunavir, tipranavir, telaprevir, saquinavir, darunavir, fosamprenavir, boceprevir, gemfibrozil, fenofibrate, etc)
* Any serious underlying medical condition (by the investigator's judgement) which could impair the ability of the patient to participate in the trial
* Patients with hereditary galactose intolerance, Lapp-lactase deficiency or Glucose-Galactose-malabsorption
* Compliance with trial medical follow-up impossible due to geographic, social or psychological reasons
* Psychiatric disorder precluding understanding of information about trial related topics, providing informed consent, or interfering with compliance for oral drug intake

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 1210 (Estimated)
Dates: Start 2019-06-06 (Actual); Primary Completion 2042-03 (Estimated); Study Completion 2042-03 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | OS will be calculated from the date of randomization to the date of death up to 15 years

CONTACTS AND LOCATIONS:
Locations (23):
- Studentova, Olomouc, Czechia
- France (11):
  - Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val De Marne
  - CHU Besançon Hopital Jean Minjoz, Besançon
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Azuréen de Cancérologie, Mougins
  - Centre Antoine Lacassagne, Nice
  - Hôpital de la Croix Saint Simon, Paris
  - Institut Jean Godinot, Reims
  - Hôpital d'Instruction des Armées Bégin, Saint-Mandé
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Hôpital Foch, Suresnes
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
- Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, Cosenza, Italy
- NOVOTNA, Bratislava, Slovakia
- Switzerland (8):
  - Klinik Hirslanden Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Bellinzona Istituto Oncologico, Bellinzona
  - Kantonsspital Baselland, Bruderholz
  - Kantansspital Graubündern, Chur
  - Kantonsspital Münsterlingen, Münsterlingen
  - Kantonsspital St.Gallen, Sankt Gallen
  - Stadtspital Triemli, Zurich
- AYADI, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided